CLINICAL TRIAL: NCT01056237
Title: Research Institute of Nephrology, Jinling Hospital,
Brief Title: Long-Term Study of Multi-target Therapy as Maintenance Treatment for Lupus Nephritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhi-Hong Liu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1002
Record Dates: First submitted 2010-01-21; First posted 2010-01-26 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-target therapy (Experimental): (Tarcrolimus+mycophenolate mofetil)
  Interventions: Drug: Multi-target therapy
- Azathioprine (Active Comparator): Aza
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Multi-target therapy — Tacrolimus (1-3mg/d) and mycophenolate mofetil(0.5-0.75g/d)
  Other Names: Tacrolimus+mycophenolate mofetil
  Arms: Multi-target therapy
Drug: Azathioprine — 1.0-2.0mg/kg/d
  Other Names: Aza
  Arms: Azathioprine

SUMMARY:
An multi-site, randomized, prospective study to compare the efficacy and safety of multi-target therapy as continuous induction and maintenance treatment versus CTX- Aza therapy.

DETAILED DESCRIPTION:
Azathioprine (AZA) has been used for maintenance therapy of lupus nephritis for many years. We compare the efficacy and safety of multi-target therapy as continuous induction and maintenance treatment vs CTX-Aza.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who signed written informed consent form
2. SLE patient, aged between 18-65 years, female or male;
3. Patients diagnosed lupus nephritis according to ISN/RPS 2003 classification criteria, class Ⅲ, Ⅳ,Ⅳ+Ⅴ, Ⅲ+Ⅴ or Ⅴ LN by renal biopsy
4. All patients had received induction therapy for 6 months with multi-therapy (FK506 + MMF) or intravenous CTX pulses.
5. Patients were recruited when received partial remission or complete remission after 6 months induction therapy.

Complete remission: proteinuria <0.4 g/24h, negative urine sediment, serum albumin >35 g/L, elevated scr <0.3mg/dl, no extra-renal complications; Partial remission: proteinuria <1.0 g/24h, urine RBC <50X104/ml without casts, serum albumin > 30 g/L, elevated Scr <0.3mg/dl,no extra-renal complications.

Exclusion Criteria:

1. Patients who didn't sign written informed consent form or could not obey the protocol.
2. Patients who didn't received the CR or PR criterion.
3. Patients who have impaired liver function, with ALT/GPT or AST/GOT twice more than the normal upper limit or who have active hepatitis.
4. WBC <3000/mm3 in peripheral blood .
5. Patients with central nervous system symptoms. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy and safety of multi-target therapy as maintenance treatment for lupus nephritis with Aza. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: zhihong Liu, Master, Principal Investigator — Research Institute of Nephrology, Jinling Hospital
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing, Jiangsu, China